CLINICAL TRIAL: NCT00758238
Title: Evidence-Based Development and Initial Evaluation of a Facilitated Patient Self Management e Health Strategy Intervention for Hypertension
Brief Title: Development and Pilot-Testing of a Patient Self Management Approach for Hypertension Using Personal Electronic Health Records
Acronym: myBP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hamilton Health Sciences Corporation (Other)
Responsible Party: Lisa Dolovich, David Chan, Tina Karwalajtys (co-principal investigators), McMaster University, Department of Family Medicine
Organization: McMaster University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 8-42213
Record Dates: First submitted 2008-09-23; First posted 2008-09-25 (Estimated); Last update posted 2008-09-25 (Estimated); Status verified 2008-09

CONDITIONS: Hypertension
Keywords: hypertension; self-management; e-health
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- myBP intervention (Experimental): participants will receive access to hypertension self-management tools and support via a personal patient electronic health record
  Interventions: Other: myBP facilitated e-health self-management
- usual care (No Intervention): participants allocated to usual care may still opt to use the personal patient electronic health record, but will not have access to the hypertension self-management tools until after the intervention period. The usual care group will be given a web-link for patient hypertension management resources

INTERVENTIONS:
Other: myBP facilitated e-health self-management — MyOSCAR, a web-based patient-controlled personal health record, provides a mechanism for patients to enter/track health information and can encourage longitudinal patient engagement, better interaction between patients and health care providers, and patient self management. The intervention will provide access via MyOSCAR to a cardiovascular risk profile and BP tracker with sharing to providers enabled. Patients can receive general information about hypertension management; tailored messages related to their modifiable risk factors; and secure messaging with multiple providers. Providers can draw on a 'menu' of links/resources to share with patients. A lifestyle changes planner/checklist and an enhanced medication diary are additional components.
  Arms: myBP intervention

SUMMARY:
The project includes a systematic review to inform refinement of intervention components and a pilot RCT to determine the uptake, feasibility, and potential value of a hypertension self-management strategy using personal health records. The review follows generally acceptable systematic review and/or meta-analytic techniques; with specific attention devoted towards accessing information and effectiveness data from unpublished studies or reports within grey literature and contacting individuals with expertise in chronic disease management in primary care. Findings of the review will be used to expand/modify an existing intervention 'template' to yield an evidence-based strategy with potential to enhance self-management of hypertension in primary care. The pilot RCT will assess the utility of the multifaceted intervention, delivered in part via a secure patient-controlled personal electronic health record, compared with the usual family practice management, for patients with undiagnosed or uncontrolled elevated blood pressure. Patients who are hypertensive or identified as high risk are expected to benefit from the increased flexibility and autonomy of out-of-physician-office self-monitoring with self-management support. This initial evaluation will focus on the change in hypertension knowledge, patient self-efficacy, and patient engagement in self management activities after 3 months, in the intervention group compared to the control group; the feasibility and acceptability of the intervention to patients and providers; and the processes involved in linking the patient self-management experience back to the patient's health care providers to promote coordination of care. Secondary outcomes include change in blood pressure, number and content of interactions with providers, and changes in management, including antihypertensive medication.

ELIGIBILITY:
Inclusion Criteria:

* Over 40 years of age
* Diagnosed with HTN, or being monitored for diagnosis, with a systolic BP >140 (SBP >130 mmHg if diabetes is diagnosed) at an office visit in the previous 6 months
* Own, borrow or be interested in purchasing a BP measurement device for home monitoring; or visit the clinic for self-assessment using the BpTRUTM (www.bptru.org)or monitor BP with a consistent device at a community pharmacy
* Regular access to email, to receive notices of new messages or prompts/reminders in MyOSCAR

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2008-09; Primary Completion 2009-06 (Estimated); Study Completion 2009-09 (Estimated)

PRIMARY OUTCOMES:
Change in hypertension knowledge, patient self-efficacy, and patient engagement in self management activities after 3 months, in the intervention group compared to the control group | 3 months

SECONDARY OUTCOMES:
Changes in blood pressure and antihypertensive medications | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Dolovich, PharmD, Principal Investigator — McMaster University; David Chan, MD, Principal Investigator — McMaster University; Tina Karwalajtys, PhD, Principal Investigator — McMaster University
Locations (1):
- Stonechurch Family Health Centre and McMaster Family Practice, Hamilton, Ontario, Canada